CLINICAL TRIAL: NCT05503225
Title: Colchicine Use in Intracranial Atherosclerotic Disease - a Pilot Open-labelled Randomized Trial
Brief Title: Colchicine Use in Intracranial Atherosclerotic Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. IP Yiu Ming Bonaventure, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CREC No. 2022.008
Record Dates: First submitted 2022-07-29; First posted 2022-08-16 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: ICAD - Intracranial Atherosclerotic Disease
Keywords: ICAD; CVA; colchicine
MeSH Terms: conditions — Intracranial Arteriosclerosis | interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: A 1:1 recruitment ratio of treatment to control group will be recruited. A sample size of 25 patients per arm will be required, therefore a total sample size of 50 will be required. Assuming a 30% rate of lost-to-follow-up, a sample size of 72 will be required.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Colchicine (Active Comparator): 0.5 mg of Colchicine for 12 months to be orally taken
  Interventions: Drug: Colchicine 0.5 MG
- Standard of care (No Intervention): Standard medical therapy

INTERVENTIONS:
Drug: Colchicine 0.5 MG — 0.5mg Orally Taken Colchicine
  Arms: Colchicine

SUMMARY:
Intracranial atherosclerotic disease (ICAD) is a major ischaemic stroke aetiology in Asia. Influenced by genetics, lifestyle and metabolic risk factors. From the SAMMPRIS cohort, 1-year stroke recurrence risk was 13% even with intensive medical therapy.

In this pilot randomized, double-blind, placebo-controlled trial, the investigators shall recruit 44 patients with recent ischaemic stroke due to intracranial atherosclerosis (ICAD) with ≥ 50% stenosis. Patients will be randomly assigned to either low-dose colchicine (0.5mg daily) (n=22) or placebo (n=22) for 12 months. High-resolution magnetic resonance vessel wall imaging will be performed at baseline and 12 months. The primary endpoint is a composite of regression of intracranial stenosis, plaque volume, or occurrence of any major adverse cardio- or cerebrovascular events at 12 months. The investigators shall also evaluate safety endpoints including diarrhea, marrow suppression, infections, neuromuscular dysfunction.

No studies had focused on the use of colchicine in patients with ICAD, which is highly prevalent in Asia. Results from this pilot trial will provide an important basis for a larger-scale main trial in the future.

DETAILED DESCRIPTION:
Background:

Intracranial atherosclerotic disease (ICAD) is a major ischaemic stroke aetiology in Asia. Influenced by genetics, lifestyle and metabolic risk factors, over 40% of ischaemic strokes were related to ICAD in China. ICAD also predicted high risk of recurrence compared to other stroke aetiologies. From the SAMMPRIS cohort, 1-year stroke recurrence risk was 13% even with intensive medical therapy. While up-front endovascular intervention resulted in unacceptably high peri-procedural stroke risk of 20%-36%, minimal advances in medical therapy targeting ICAD had been made.

Literature clinical findings were supported by coronary plaque-imaging studies performed in human and animal models, which showed coronary plaque regression in patients with recent acute coronary syndrome and reduction in abdominal-aortic plaque inflammation in a rabbit-model. In parallel, under intensive medical therapy, ICAD plaque regression could be seen in 49% of patients. Nevertheless, recurrent stroke rate still exceeded 10% despite treatment targets of blood pressure ≤140/90, HbA1c ≤6.5%, and low-density lipoprotein (LDL) ≤1.8mmol/L in our previous cohort. There is a need to further reduce plaque growth, thrombogenicity and haemodynamic compromise by intensifying anti-atherosclerotic therapy. An updated meta-analysis showed that colchicine use in patients with high cardiovascular risk was associated with lower stroke incidence (12). However, no studies had focused on the use of colchicine in patients with ICAD, which is highly prevalent in Asia.

Objective:

In this pilot randomized, double-blind, placebo-controlled trial, the investigators aim to elucidate the efficacy and safety of low-dose colchicine (0.5mg daily) in patients with symptomatic intracranial atherosclerotic disease. The investigators hypothesize that low-dose colchicine in addition to intensive medical therapy, compared to intensive medical therapy alone, may result in more plaque regression in patients with symptomatic ICAD. Results from this pilot trial will provide an important basis for a larger-scale main trial in the future.

Methods:

In this pilot randomized, double-blind, placebo-controlled trial, the investigators shall recruit 44 patients with recent ischaemic stroke due to intracranial atherosclerosis (ICAD) with ≥ 50% stenosis. Patients will be randomly assigned to either low-dose colchicine (0.5mg daily) (n=22) or placebo (n=22) for 12 months. High-resolution magnetic resonance vessel wall imaging will be performed at baseline and 12 months. The primary endpoint is a composite of regression of intracranial stenosis, plaque volume, or occurrence of any major adverse cardio- or cerebrovascular events at 12 months. The investigators shall also evaluate safety endpoints including diarrhea, marrow suppression, infections, neuromuscular dysfunction.

Significance:

No studies had focused on the use of colchicine in patients with ICAD, which is highly prevalent in Asia. Results from this pilot trial will provide an important basis for a larger-scale main trial in the future.

ELIGIBILITY:
Inclusion Criteria

1. Chinese patients aged 40-80 years old
2. Patients with symptomatic ICAD of ≥ 50% stenosis in middle cerebral arteries, basilar artery. Degree of stenosis will be quantified by computer tomographic angiography (CTA), magnetic resonance imaging (MRI) or digital subtraction angiography (DSA) by the WASID method (13). Symptomatic ICAD is defined as ischemic stroke or transient ischemic attack with clinical or radiological signs correspond to the vascular territory supplied by the disease vessel.
3. Patients with first-ever ischaemic stroke within 8 weeks of recruitment

Exclusion Criteria

1. Patients who are unable to provide an informed consent
2. Patients who are contraindicated to contrast MRI scans, e.g. non-MRI compatible pacemaker, claustrophobia, known gadolinium-based contrast allergy, estimated glomerular filtration rate < 30mL/min/1.73m2, etc.
3. Patients who have absolute or relative contraindications to colchicine therapy, e.g. colchicine allergy, neuromuscular disorders, haematological diseases, chronic diarrhea, estimated glomerular filtration rate < 30mL/min/1.73m2, chronic liver disease, etc.
4. Patients with intracranial stenosis not due to atherosclerosis, e.g. vasculitis, vasospasm, Moyamoya disease, etc.
5. Pregnancy
6. Patients with elevated creatine kinase level at randomisation stage of study.
7. Recurrent gouty arthritis that requires colchicine for > 3 months per year;
8. Inflammatory bowel disease or chronic diarrhea;
9. Neuromuscular disease or a nontransient creatine kinase level that was greater than three times the upper limit of the normal range (unless due to infarction) for > 3 months;
10. Clinically significant nontransient hematologic abnormalities with hemoglobin <10g/dL, white blood cell < 4x10^9, or platelet < 100x10^9/L for > 3 months;
11. Alcoholism;
12. Long term systemic glucocorticoid therapy

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-11-28 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Regression of intracranial stenosis | at 12 months
  Regression in stenosis of ≥ 15% using the WASID method.
Regression of plaque volume | at 12 months
  Regression of plaque burden of ≥ 15% compared to baseline.
Major adverse cardio- or cerebrovascular events (MACE) | at 12 months
  Occurrence of any major adverse cardio- or cerebrovascular events (MACE).

SECONDARY OUTCOMES:
Longitudinal changes in ICAD stenosis | at 12 months
  Subjects will receive a novel high-resolution magnetic resonant vessel-wall imaging which depicts the degree of symptomatic stenosis, plaque burden, plaque enhancement, plaque remodelling and intraplaque haemorrhage.
Longitudinal changes in plaque volume | at 1,3,6,9,12 months
  Longitudinal changes in plaque volume by DSA or equivalent imaging techniques.
Longitudinal changes in resolution of plaque enhancement | at 1,3,6,9,12 months
  Longitudinal changes in resolution of plaque enhancement by DSA or equivalent imaging techniques.
Longitudinal changes in white matter hyperintensity volume | at 12 months
  Longitudinal changes in white matter hyperintensity volume by MRI or equivalent imaging.
Longitudinal changes in number of silent lacunes | at 12 months
  Longitudinal changes in number of silent lacunes by MRI or equivalent imaging.
Longitudinal changes in cognitive ability | at 1,3,6,9,12 months
  Longitudinal changes in cognitive ability by assessment: Hong Kong Montreal Cognitive Assessment (5-min Protocol).

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No